CLINICAL TRIAL: NCT04236102
Title: Use of the Biocartis Idylla ™ Platform for the Detection of Epidermal Growth Factor Receptor, B-RAF and K-RAS Proto-oncogene Mutations in Liquid Based Cytology Specimens and Blood Plasma Samples From Patients With Non Small Cell Lung Carcinoma and Pancreatic Adenocarcinoma
Brief Title: KEBI-Cyto Study - Use of the Biocartis Idylla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Cornwall Hospitals Trust (Other)
Collaborators: Biocartis NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019.RCHT.111
Record Dates: First submitted 2020-01-10; First posted 2020-01-22 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Adenocarcinoma; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Genes, ras

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EGFR, KRAS, BRAF Lung adenocarcinoma LBC (Experimental): Will use residual material from existing LBC cytology samples sent to the laboratory. Routine testing will take priority. Cases identified as non small cell lung carcinoma will have the residual LBC sample tested on the Idylla platform for EGFR, KRAS and BRAF. The EGFR, KRAS and BRAF mutation results obtained using the routine diagnostic procedure (FFPE samples) will be compared to those produced using the LBC samples.
  Interventions: Diagnostic Test: Biocartis Idylla platform - real time PCR detecting EGFR, KRAS and BRAF mutations in liquid based cytology and blood plasma samples
- KRAS Pancreatic adenocarcinoma (Experimental): Will involve testing archived FFPE clot samples from confirmed pancreatic adenocarcinoma patients since 2014 (Approximately 20 cases per year). KRAS testing will be performed using the Idylla platform to establish if there is a KRAS codon 12 mutation present in 94% percent of the cases reported at RCHT. Patients will have consented to the use of their tissue at the time of procedure. Prospectively new patients diagnosed with pancreatic adenocarcinoma will have KRAS testing on the FFPE clot made as part of the routine diagnostic work up and KRAS testing on the LBC sample.
  Interventions: Diagnostic Test: Biocartis Idylla platform - real time PCR detecting EGFR, KRAS and BRAF mutations in liquid based cytology and blood plasma samples
- EGFR, KRAS, BRAF Blood plasma (Experimental): Will involve a blood sample being taken at the time of the procedure from patients that have a clinical suspicion of having lung or pancreatic cancer. The single blood sample will be taken from the cannula inserted for the procedure. The blood sample will be processed using the Biocartis Idylla ™ circulating tumour cell cartridges (EFGR, KRAS and BRAF for lung and KRAS for pancreas).
  Interventions: Diagnostic Test: Biocartis Idylla platform - real time PCR detecting EGFR, KRAS and BRAF mutations in liquid based cytology and blood plasma samples

INTERVENTIONS:
Diagnostic Test: Biocartis Idylla platform - real time PCR detecting EGFR, KRAS and BRAF mutations in liquid based cytology and blood plasma samples — Automated real time PCR mutation analysis - 1. Can the Idylla platform provide a standardised and effective method for detecting EGFR, KRAS and BRAF mutations in blood and liquid based cytology samples for patients with lung and pancreatic cancer. Mutation detection increases the treatment options for patients.

SUMMARY:
Use of the Biocartis Idylla ™ platform for the detection of Epidermal Growth Factor Receptor, B-RAF and K-RAS proto-oncogene mutations in liquid based cytology specimens and blood plasma samples from patients with non small cell lung carcinoma and pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Advances in medicine have resulted in the development of specific drugs to treat cancers that express certain mutations. The detection of epidermal growth factor receptor (EGFR), BRAF and KRAS mutations (10-30%, 1-2%, 25% respectively) in lung cancers and KRAS mutations in 94% of pancreatic cancers allows these patients to be treated with a wider cohort of drugs, potentially resulting in progression free, prolonged survival, with a more favourable tolerability and less adverse effects compared with chemotherapy.

NHS England has a test directory which lists the molecular tests that trusts should provide for cancer patients. EGRF, KRAS and BRAF are listed in this directory. Verification of the use of the Idylla would enable this trust to provide all of these molecular tests effectively. Lung and pancreatic cancers both present at advanced disease states and therefore a rapid turnaround of test results is vital. Currently laboratories rely on the use of formalin-fixed paraffin embedded (FFPE) samples for EGFR testing.

Clots are produced in the laboratory to congeal all of the tissue fragments and cells into one solid mass. The clotted sample is then fixed in formalin and processed. The current processing and reporting time is 5 days. Liquid based cytology (LBC) specimens obtained through the same sampling procedures are also prepared in the laboratory and fixed using a methanol based fixative called Preservcyt. Previous research has been conducted to determine whether LBC samples can be used instead of FFPE samples for mutation detection with favourable results. A switch to the use of LBC samples for mutation analysis on the Idylla would remove multiple processing steps and make use of residual samples that are currently discarded, which optimises the amount of testing that we can run on small cytology samples, reducing the likelihood of repeat procedures for patients. Alcohol fixation is regarded as a superior method of DNA and RNA preservation, therefore better molecular results will be seen.

Detection of circulating tumour cell mutations could in the future negate the need for invasive procedures, with patients requiring a simple blood test for diagnosis.

The aim of the study is to determine whether LBC samples are a feasible and reliable alternative to FFPE samples for detecting mutations in LBC samples and blood using the Idylla platform.

Hypothesis: EFGR, KRAS and BRAF mutations identified using FFPE samples will be detected in LBC and blood plasma samples using the Biocartis Idylla ™ platform.

Part 1 of the study: (extension of previous research project - IRAS Number: 261622) Will use residual material from existing LBC cytology samples sent to the laboratory. Routine testing will take priority. Cases identified as non small cell lung carcinoma will have the residual LBC sample tested on the Idylla platform for EGFR, KRAS and BRAF. The EGFR, KRAS and BRAF mutation results obtained using the routine diagnostic procedure (FFPE samples) will be compared to those produced using the LBC samples.

Part 2 of this study:

Will involve testing archived FFPE clot samples from confirmed pancreatic adenocarcinoma patients since 2014 (Approximately 20 cases per year). KRAS testing will be performed using the Idylla platform to establish if there is a KRAS codon 12 mutation present in 94% percent of the cases reported at RCHT. Patients will have consented to the use of their tissue at the time of procedure. Prospectively new patients diagnosed with pancreatic adenocarcinoma will have KRAS testing on the FFPE clot made as part of the routine diagnostic work up and KRAS testing on the LBC sample.

Part 3 of this study:

Will involve a blood sample being taken at the time of the procedure from patients that have a clinical suspicion of having lung or pancreatic cancer. The single blood sample will be taken from the cannula inserted for the procedure. The blood sample will be processed using the Biocartis Idylla ™ circulating tumour cell cartridges (EFGR, KRAS and BRAF for lung and KRAS for pancreas).

Samples for inclusion in the study will be identified by a (member of direct care team) working in the cytology department who will perform a computerised search every week and identify patients who have been diagnosed with non small cell lung carcinoma or pancreatic adenocarcinoma. The patient's original laboratory number will be entered into a secure, password protected database and the patient will then be assigned with a new study number. This database, and patient information, will only be accessible by the senior biomedical scientist and will be stored in a secure electronic file in compliance with information governance and patient confidentiality. Patient samples will be labelled with the study number and the original laboratory number and all patient information will be covered. The researcher will not have access to any patient information and will not be able to identify any patients. The senior biomedical scientist will store the anonymised results of the study into the database. The study duration will be 24 months. In which time it is estimated that the following number of patients will be tested:

100 patients for non small cell lung carcinoma 60 retrospective pancreatic adenocarcinoma samples 40 prospective pancreatic adenocarcinoma patients

Patients attending for EUS (Endoscopic ultrasound) or EBUS (Endobronchial ultrasound) guided fine needle aspirations with a clinical suspicion of non-small cell lung carcinoma or pancreatic carcinoma by multi-disciplinary team. Samples for inclusion in the study will be identified by a senior biomedical scientist (member of direct care team) working in the cytology department who will perform a computerised search every week and identify patients who have been diagnosed with lung non-small cell carcinoma and pancreatic adenocarcinoma. The patient's original laboratory number will be entered into a secure, password protected database and the patient will then be assigned with a new study number. This database, and patient information, will only be accessible by the senior biomedical scientist and will be stored in a secure file in compliance with information governance and patient confidentiality. Patient samples will be labelled with the study number and the original laboratory number and all patient information will be covered. The researcher will not have access to any patient information and will not be able to identify any patients. Samples that do not meet the study criteria will be discarded in accordance with laboratory protocol.

All patient data (including tissue samples and associated reports) will be anonymised prior to being released to the primary researcher. The identifiable data is linked by a laboratory number. This information is stored in a secure database accessible only by a member of the direct care team.

All information is stored and backed up on secure servers at the Royal Cornwall Hospital. All databases relevant to the research will be password protected and this is monitored by the RCHT IT department. The location of the databases themselves will only be accessible to authorised users.

No further patient intervention is required for this research.

If liquid based cytology (LBC) samples are found to be a feasible alternative for EGFR, KRAS and BRAF mutation testing this has the potential to result in:

* Quicker turnaround time of results in cases of unequivocal adenocarcinoma. This would provide
* Earlier access to treatment allowing for optimal patient management.
* Expands the range of molecular testing provided in house as recommended by the NHS test library.
* Easier sample preparation within the laboratory
* Increase in efficient use of material could also prevent repeat sampling procedures on patients.
* Use of LBC samples may allow for better results from molecular testing (methanol superior fixative to formalin).
* Supports of the use of blood sample testing for circulating tumour cells (less invasive sampling). This may identify at what disease staging circulating tumour cells can be detected in blood plasma, which would make it a potential future diagnostic triaging and follow up tool.
* Supports KRAS mutation testing for pancreatic adenocarcinoma and future development of target therapies specific to the codon 12 mutation

ELIGIBILITY:
Inclusion Criteria:

* Cytological / histological diagnosis of non small cell lung carcinoma or pancreatic adenocarcinoma
* Patients of any gender ethnicity or socioeconomic grouping
* Patients over the age of 18 years

Exclusion Criteria:

* Other malignancies (Not non small cell lung carcinoma or pancreatic adenocarcinoma)
* Benign diagnosis
* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
The number of participants with negative and positive mutation status for KRAS, EGFR and BRAF in LBC samples detected using the BioCartis Idylla Platform real time PCR kits. | 24 months
  1. Can the Idylla platform provide a standardised and effective method for detecting EGFR, KRAS and BRAF mutations in liquid based cytology samples for patients with lung and pancreatic cancer. Mutation detection increases the treatment options for patients.
The number of patients with a positive KRAS mutation status in Cytolgy clot samples reported as pancreatic adenocarcinoma, using the Biocartis Idylla platform real time PCR kits. | 24 months
  2. Establish the mutation prevalence in population served by the Royal Cornwall Hospital. This could provide an avenue for drug development to treat pancreatic cancers
The number of participants with negative and positive mutation status for KRAS, EGFR and BRAF in blood plasma samples detected using the BioCartis Idylla Platform real time PCR kits. | 24 months
  3. Testing for mutations in the blood samples and directly comparing it with mutations seen in the cytology samples, will provide valuable information in the reliance of blood tests for cancer diagnosis. Potentially eliminating the need for invasive procedures in the future.

CONTACTS AND LOCATIONS:
Overall Officials: James Garvican, Principal Investigator — Royal Cornwall Hospitals Trust
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao H, Qiu T, Guo H, Ying J, Li J, Zhang Z. Detection of EGFR and KRAS gene mutations using suspension liquid-based cytology specimens in metastatic lung adenocarcinoma. Oncotarget. 2017 Nov 20;8(63):106685-106692. doi: 10.18632/oncotarget.22530. eCollection 2017 Dec 5. PMID 29290981
- [Result] De Luca C, Gragnano G, Pisapia P, Vigliar E, Malapelle U, Bellevicine C, Troncone G. EGFR mutation detection on lung cancer cytological specimens by the novel fully automated PCR-based Idylla EGFR Mutation Assay. J Clin Pathol. 2017 Apr;70(4):295-300. doi: 10.1136/jclinpath-2016-203989. Epub 2016 Aug 19. PMID 27543600
- [Result] Hadano N, Murakami Y, Uemura K, Hashimoto Y, Kondo N, Nakagawa N, Sueda T, Hiyama E. Prognostic value of circulating tumour DNA in patients undergoing curative resection for pancreatic cancer. Br J Cancer. 2016 Jun 28;115(1):59-65. doi: 10.1038/bjc.2016.175. Epub 2016 Jun 9. PMID 27280632
- [Result] Sausen M, Phallen J, Adleff V, Jones S, Leary RJ, Barrett MT, Anagnostou V, Parpart-Li S, Murphy D, Kay Li Q, Hruban CA, Scharpf R, White JR, O'Dwyer PJ, Allen PJ, Eshleman JR, Thompson CB, Klimstra DS, Linehan DC, Maitra A, Hruban RH, Diaz LA Jr, Von Hoff DD, Johansen JS, Drebin JA, Velculescu VE. Clinical implications of genomic alterations in the tumour and circulation of pancreatic cancer patients. Nat Commun. 2015 Jul 7;6:7686. doi: 10.1038/ncomms8686. PMID 26154128